CLINICAL TRIAL: NCT04075162
Title: Community Benefit of No-charge Calcium Score Screening Program
Acronym: CLARIFY
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Sanjay Rajagopalan, Division Chief of Cardiovascular Medicine, University Hospitals Cleveland Medical Center
Other Study IDs: 20190995
Record Dates: First submitted 2019-08-21; First posted 2019-08-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low charge CAC: Patients receiving CAC for Cardiovascular disease risk screening at low charge (99 USD)
- No charge CAC: Patients receiving CAC for Cardiovascular disease risk screening at no charge

SUMMARY:
Current approaches in primary prevention for cardiovascular disease are based on probabilistic approaches to estimate risk, using many of the widely available cardiovascular risks scores, with over 100 such scoring systems currently available throughout the world. The rationale for this practice is to select those individuals at greatest risk for more intense targets, reduce risk of treatment to those at minimal risk, and to maximize the cost-effectiveness of treatment. A recent Cochrane Systematic Review assessed the practice of using risk scores to select individuals for the primary prevention of cardiovascular disease. 3 The principal finding of the systematic review was that there was little or no effect of providing clinicians with cardiovascular risk scores when compared to standard of care (5.4% versus 5.3%; relative risk 1.01, 95% confidence intervals 0.95 to 1.08). The authors concluded that there is major uncertainty whether current strategies for providing risk scores and called for further research to address this concern. Extent of coronary artery calcium (CAC) is a strong risk marker for coronary events, with evidence mainly derived from observational studies and from prospective non-randomized studies. CAC, although endorsed for intermediate risk patients, is not widely adopted due to barriers in reimbursement. The cost of the test ranges between 100 and 300 USD in the United States, which may have limited the wide adoption of the test. Whether reducing the cost burden for CAC increases utilization for routine screening and its influence on physician practices and downstream testing is largely unknown. University Hospitals started offering low charge CAC (99$) since 2014. In 2017, University Hospitals started offering CAC for no charge for patients to improve access to this test, which has not traditionally been covered by insurance companies. The impact of no-charge CAC has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Received Coronary Artery Calcium (CAC) CT scan at University Hospitals starting in January 1, 2014.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who received a no-cost Coronary Artery Calcium (CAC) CT scan at University Hospitals (Cleveland, Oh) starting in January 1, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 77000 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Statin Prescription | 1 year

SECONDARY OUTCOMES:
Non-invasive coronary ischemia testing | 1 year
  Stress echocardiograms, myocardial perfusion imaging
Invasive coronary ischemia testing | 1 year
  Invasive coronary angiography
Coronary revascularization procedures | 1 year
  Percutaneous coronary interventions, coronary artery bypass grafting

OTHER OUTCOMES:
LDL cholesterol | 1 year
  Change in LDL cholesterol levels from baseline to 1 year
Total cholesterol | 1 year
  Change in LDL cholesterol levels from baseline to 1 year
Blood pressure | 1 year
  Change in blood pressure from baseline to 1 year
Body mass index | 1 year
  Change in BMI from baseline to 1 year
Serum Triglycerides | 1 year
  Change in BMI from baseline to 1 year
Myocardial infarction | 1 year
  Incidence of myocardial infarction
Stroke | 1 year
  Incidence of myocardial infarction
Death | 1 year
  Incidence of death
Lung cancer | 1 year
  Incidence of lung cancer

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Singh P, Hoori A, Freeze J, Hu T, Tashtish N, Gilkeson R, Li S, Rajagopalan S, Wilson DL, Al-Kindi S. Leveraging calcium score CT radiomics for heart failure risk prediction. Sci Rep. 2024 Nov 6;14(1):26898. doi: 10.1038/s41598-024-77269-x. PMID 39505933
- [Derived] Hoori A, Al-Kindi S, Hu T, Song Y, Wu H, Lee J, Tashtish N, Fu P, Gilkeson R, Rajagopalan S, Wilson DL. Enhancing cardiovascular risk prediction through AI-enabled calcium-omics. Sci Rep. 2024 May 15;14(1):11134. doi: 10.1038/s41598-024-60584-8. PMID 38750142
- [Derived] Hoori A, Al-Kindi S, Hu T, Song Y, Wu H, Lee J, Tashtish N, Fu P, Gilkeson R, Ra-Jagopalan S, Wilson DL. Enhancing cardiovascular risk prediction through AI-enabled calcium-omics. ArXiv [Preprint]. 2023 Aug 23:arXiv:2308.12224v1. PMID 37664409
- [Derived] Siva Kumar S, Al-Kindi S, Tashtish N, Rajagopalan V, Fu P, Rajagopalan S, Madabhushi A. Machine learning derived ECG risk score improves cardiovascular risk assessment in conjunction with coronary artery calcium scoring. Front Cardiovasc Med. 2022 Oct 5;9:976769. doi: 10.3389/fcvm.2022.976769. eCollection 2022. PMID 36277775
- [Derived] Al-Kindi S, Tashtish N, Rashid I, Sullivan C, Neeland IJ, Robinson M, Gross EM, Shaw L, Cainzos-Achirica M, Nasir K, Kreatsoulas C, Gilkeson R, Simon DI, Rajagopalan S. Impact of low/no-charge coronary artery calcium scoring on statin eligibility and outcomes in women: The CLARIFY study. Am J Prev Cardiol. 2022 Sep 11;12:100392. doi: 10.1016/j.ajpc.2022.100392. eCollection 2022 Dec. PMID 36157553
- [Derived] Khawaja T, Janus SE, Tashtish N, Janko M, Baeza C, Gilkeson R, Al-Kindi SG, Rajagopalan S. Prevalence of thoracic aortic aneurysm in patients referred for no/low-charge coronary artery calcium scoring: Insights from the CLARIFY registry. Am J Prev Cardiol. 2022 Aug 30;12:100378. doi: 10.1016/j.ajpc.2022.100378. eCollection 2022 Dec. PMID 36106308